CLINICAL TRIAL: NCT07117305
Title: A Clinical Investigation Into the Safety and Efficacy of CD7 Chimeric Antigen Receptor T-cell (CAR-T) Therapy in Combination With Autologous Hematopoietic Stem Cell Transplantation for the Treatment of Relapsed/Refractory T-cell Lymphoma
Brief Title: CD7 CAR-T Combined With Autologous Hematopoietic Stem Cell Transplantation
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhengzhou University (Other)
Collaborators: Hebei Taihe Chunyu Biotechnology Co., Ltd (Industry)
Responsible Party: Principal Investigator, Mingzhi Zhang, the director of oncology department of the first affiliated hospital Investigator Affiliation, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-Th-C252-V1.0
Record Dates: First submitted 2025-06-18; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: CD7+ Lymphoma; T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD7+ T cell lymphoma (Experimental)
  Interventions: Drug: CD7 CAR-T combined with autologous hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: CD7 CAR-T combined with autologous hematopoietic stem cell transplantation — Phase I adopts a standard 3+3 dose-escalation design (with exploratory doses of 1×10⁶, 2×10⁶, and 2.5×10⁶ CAR⁺ cells/kg) to determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D). Phase II expands at the RP2D to further assess efficacy.
  During screening, eligible patients will be identified and consented. In the collection phase, patients undergo two separate apheresis procedures: G-CSF-mobilized peripheral blood stem cell collection for ASCT and PBMC collection for CAR-T manufacturing. Bridging therapy and gut preparation may be performed. The pretreatment phase(recommended: BEAM therapy) starts from Day -8. Investigators may adjust the pretreatment regimen based on the patient's performance. On Day 0, autologous stem cells are infused. CD7 CAR-T cells are infused on Days 2-7 post-transplant. Follow-up visits occur on Days 10, 14, 21, 28, and Months 2, 3, 6, and 12.

SUMMARY:
This is a single-arm, open-label, phase I/II clinical trial initiated by investigators to evaluate the safety, tolerability, and preliminary efficacy of CD7-targeted chimeric antigen receptor T cells (CD7 CAR-T) combined with autologous stem cell transplantation (ASCT) in patients with relapsed or refractory CD7-positive T-cell lymphomas. Phase I adopts a standard 3+3 dose-escalation design to determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D). Phase II expands at the RP2D to further assess efficacy. The study includes lymphodepletion chemotherapy, ASCT, and sequential infusion of CD7 CAR-T cells. The primary objectives include: (1) Evaluate safety/tolerability of CD7 CAR-T + auto-HSCT in relapsed or refractory CD7-positive T-cell lymphomas. (2) Determine MTD and RP2D. The secondary objectives include: (1) Assess efficacy (overall response rate, complete response, duration of response, progression-free survival and overall survival. (2)Characterize PK/PD profiles. (3)Investigate anti-tumor mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. With the patient's explicit consent and after signing the informed consent form, the patient is willing and capable of complying with the planned visits, research treatments, laboratory tests and other trial procedures;
2. Age range: 14 to 65 years old. Both men and women are eligible;
3. All types of CD7+ T-cell non-Hodgkin's lymphomas (except T-lymphoblastic lymphoma) diagnosed according to the World Health Organization's classification of hematopoietic and lymphoid tissue tumors (2022);
4. For patients with T-cell lymphoma who are refractory to the first-line chemotherapy regimen or who experience recurrence and resistance after at least the second-line chemotherapy regimen. The following criteria must be met: a. For those patients who had only received first-line treatment previously, if they did not achieve PR after at least 4 cycles of the first-line regimen, or if they did not achieve CR after at least 6 cycles of the first-line regimen; b. Those who experienced recurrence in the early stage (< 12 months) after complete remission; or those who experienced recurrence in the late stage (≥ 12 months) and did not achieve remission after one course of standard induction chemotherapy; c. Those who have not achieved remission after treatment with second-line or more chemotherapy regimens;
5. During the enrollment screening process, the subjects were confirmed to have CD7+ (with CD7 expression ≥ 10%) through pathological histology and/or cytology;
6. Having measurable or evaluable lesions: The target lesion is defined as a lesion within lymph nodes with a long diameter of ≥ 15mm, or an extranodal lesion larger than 10mm (in accordance with the Lugano 2014 criteria); Lesions that have received prior radiotherapy are considered measurable only if there is a clear progression after completing radiotherapy; or PET-positive lesions determined according to the Lugano criteria;
7. The Eastern Cooperative Oncology Group (ECOG) performance status score is 0 to 2, and the estimated survival period is greater than 3 months;
8. Having appropriate organ functions: a. The levels of alanine aminotransferase (ALT) and aspartate aminotransferase (AST) should be ≤ 3 times the upper limit of normal (ULN). If the abnormality of ALT and AST is judged to be caused by the disease (such as liver infiltration or bile duct obstruction), the thresholds can be relaxed to ≤ 5 times ULN; b. Total serum bilirubin ≤ 2 times ULN, except in cases where Gilbert syndrome is present; patients with Gilbert syndrome whose total bilirubin is ≤ 3 times ULN and direct bilirubin is ≤ 1.5 times ULN can be included; c. Serum creatinine ≤ 1.5 times the upper limit of normal, or creatinine clearance rate ≥ 60 mL/min; d. The international normalized ratio (INR) is no more than 1.5 times the upper limit of normal (ULN), and the activated partial thromboplastin time (aPTT) is no more than 1.5 times the ULN; e. Having the lowest level of lung reserve, defined as ≤ grade 1 dyspnea (CTCAE v5.0) and a blood oxygen saturation of ≥ 92% in the absence of oxygen supplementation; f. Left ventricular ejection fraction in echocardiography is ≥ 50%; no clinically significant abnormal electrocardiogram findings; no clinically significant pericardial effusion or pleural effusion.
9. Female participants of childbearing potential must have negative blood/urine pregnancy tests within 7 days prior to infusion. All sexually active males and females with reproductive capacity must agree to use highly effective contraception throughout the study and for at least 2 years after administration of the investigational treatment.

Exclusion Criteria:

1. Severe cardiac insufficiency with left ventricular ejection fraction (LVEF) <50%；
2. Documented history of severe pulmonary impairment；
3. History of organ transplantation or active graft-versus-host disease (GVHD);
4. Concurrent other progressive malignancies;
5. Uncontrolled severe infections;
6. Severe autoimmune diseases or primary immunodeficiency disorders;
7. Positive for any of the following: Hepatitis B surface antigen (HBsAg) and/or hepatitis B e antigen (HBeAg); Hepatitis B e antibody (HBe-Ab) and/or hepatitis B core antibody (HBc-Ab) with HBV-DNA levels above the upper limit of normal (ULN); Hepatitis C virus antibody (HCV-Ab) with detectable HCV RNA; Human immunodeficiency virus antibody (HIV-Ab); Treponema pallidum antibody (TP-Ab); Cytomegalovirus (CMV) DNA above ULN; Epstein-Barr virus (EBV) DNA above ULN；
8. History of severe hypersensitivity to biological products (including antibiotics);
9. Pre-existing central nervous system disorders, including but not limited to:

   Uncontrolled epilepsy；Cerebral ischemia/hemorrhage；Dementia；Cerebellar disorders；
10. Previous recipients of autologous or allogeneic hematopoietic stem cell transplantation;
11. Any other severe physical or psychiatric conditions or significant laboratory abnormalities that may: Increase study participation risks；Interfere with study results interpretation; Be deemed by investigators to render the patient unsuitable for study participation;
12. Presence of lymphoma-related clinical emergencies requiring immediate intervention at screening due to tumor mass obstruction or compression (e.g., intestinal obstruction, vascular compression, etc.).

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
The safety of CD7 CAR-T cell injection combined with autologous hematopoietic stem cell transplantation | Day 28 after treatment
  The possible adverse reactions recorded in each item were evaluated.

SECONDARY OUTCOMES:
Efficacy indicators | Day 28, Month 2, Month 3, Month 6, Month 12 after treatment
  The objective response rates (ORR)
Efficacy indicators | Day 28, Month 2, Month 3, Month 6, Month 12 after treatment
  The overall survival (OS)
Efficacy indicators | Day 28, Month 2, Month 3, Month 6, Month 12 after treatment
  The progression-free survival (PFS)
Efficacy indicators | Day 28, Month 2, Month 3, Month 6, Month 12 after treatment
  Complete remission (CR)
Efficacy indicators | Day 28, Month 2, Month 3, Month 6, Month 12 after treatment
  Event-free survival (EFS)
Efficacy indicators | Day 28, Month 2, Month 3, Month 6, Month 12 after treatment
  Disease Control Rate (DOCR)
kinetics of CAR-T cells | Day 28, Month 2, Month 3, Month 6, Month 12 after treatment
  Use flow cytometry or Q-PCR to monitor the kinetics of CAR-T cells.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Department of Oncology, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No